CLINICAL TRIAL: NCT00709124
Title: Use of Neuromuscular Electrostimulation (NMES) for Treatment or Prevention of ICU-Associated Weakness
Acronym: NMES
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: NA_00017423
Record Dates: First submitted 2008-07-01; First posted 2008-07-03 (Estimated); Results first posted 2015-04-16 (Estimated); Last update posted 2018-01-23 (Actual); Status verified 2018-01

CONDITIONS: Intensive Care Unit; Muscle Weakness
Keywords: Respiration, Artificial; Critical Illness; Intensive Care Units; Electric Stimulation Therapy; Muscle Weakness; Paresis; Mechanically; Ventilated; Patients; Admitted; Medical
MeSH Terms: conditions — Muscle Weakness; Respiratory Aspiration; Critical Illness; Paresis

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- NMES (Experimental): 60 minute daily NMES sessions every day for the duration of subject's ICU stay.
  Interventions: Device: Neuromuscular Electrostimulation (NMES) CareStim Muscle Stimulation Device (Care Rehab; McLean, VA)
- Sham (Sham Comparator): 60 minute sham sessions every day for the duration of subjects ICU stay. No voltage will be applied to those receiving sham sessions.
  Interventions: Device: Sham

INTERVENTIONS:
Device: Neuromuscular Electrostimulation (NMES) CareStim Muscle Stimulation Device (Care Rehab; McLean, VA) — 60 minute NMES sessions will be applied to three muscle groups of the lower extremities (quadriceps, pretibial, and triceps surae). Sessions start at study entry, and will occur every day for the duration of subject's ICU stay.
  Other Names: CareStim Muscle Stimulation Device (Care Rehab; McLean, VA)
  Arms: NMES
Device: Sham — 60 minute NMES sessions will be applied to three muscle groups of the lower extremities (quadriceps, pretibial, and triceps surae). Sessions start at study entry, and will occur every day for the duration of subject's ICU stay. Sham groups will NOT have voltage applied.
  Other Names: CareStim Muscle Stimulation Device (Care Rehab; McLean, VA)
  Arms: Sham

SUMMARY:
The purpose of this study is to investigate whether neuromuscular electrostimulation (NMES) will decrease ICU-associated weakness. The investigators believe that 60 minutes of daily NMES will improve strength and function in those who have had extended ICU stays, as well as decrease critical illness myopathy as an etiology of weakness in the critically ill.

DETAILED DESCRIPTION:
Survivors of critical illness frequently have significant, debilitating and persistent weakness after discharge from the intensive care unit (ICU). This weakness can persist for up to 4 years after ICU discharge. There are few interventions that have been successful in reducing or preventing weakness. Neuromuscular electrostimulation (NMES) therapy is beneficial in other populations of weak and functionally limited patients, such as those with chronic respiratory failure requiring mechanical ventilation, severe chronic obstructive pulmonary disease and end-stage congestive heart failure. We propose a randomized clinical trial to evaluate the efficacy of 60 minutes of NMES versus sham therapy, applied to the bilateral lower extremities, to reduce ICU-associated weakness in patients with acute respiratory failure. Our specific aims are to determine if NMES therapy will: 1) increase strength of the 3 treated lower extremity muscle groups (i.e., pretibial, triceps surae, and quadriceps), 2) improve important clinical outcomes (i.e., functional status, duration of mechanical ventilation, length of ICU and hospital stay, in-hospital mortality, and total hospital charges), 3) reduce critical illness myopathy as an etiology of weakness in clinically weak ICU patients. The investigators hypothesize that NMES therapy will reduce ICU-associated weakness, and improve clinical and functional outcomes. Additionally, the rates of critical illness myopathy as an etiology of weakness in clinically weak ICU patients will be lower in those receiving NMES versus sham therapy. Since there is no single test that is optimal for measuring muscle strength in the critically ill, the investigators will employ four non-invasive measures: manual muscle testing (MMT), hand held dynamometry (HHD), handgrip dynamometry (HGD), and maximal inspiratory pressure (MIP). With no existing therapeutic options available, our study explores the potential of NMES as a feasible intervention to reduce ICU-associated weakness.

ELIGIBILITY:
Inclusion Criteria:

* 1 day of mechanical ventilation with an expectation of requiring ≥2 additional days of ICU stay in a Johns Hopkins Intensive Care Unit (ICU)

Exclusion Criteria:

* Unable to understand or speak English due to language barrier or cognitive impairment prior to admission
* Unable to independently transfer from bed to chair at baseline prior to hospital admission
* Known primary systemic neuromuscular disease (e.g. Guillian-Barre) at ICU admission
* Known intracranial process that is associated with localizing weakness (e.g. cerebral vascular accident) at ICU admission
* Transferred from another ICU outside of the Johns Hopkins system after >4 consecutive days of mechanical ventilation
* Moribund (i.e. >90% probability of patient mortality in the next 96 hours)
* Anticipated transfer to another ICU for care (e.g. awaiting organ transplantation and transfer to surgical ICU)
* Any pacemaker (e.g., cardiac, diaphragm) or implanted cardiac defibrillator
* Pregnancy
* Body mass index ≥35 kg/m2
* Any limitation in life support other than a sole no-CPR order
* Known or suspected malignancy in the legs
* Unable to treat or evaluate both lower extremities (e.g., bilateral amputation, bilateral skin lesions)
* ICU length of stay >7 days prior to enrollment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2008-06; Primary Completion 2013-04 (Actual); Study Completion 2013-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Dale Needham, MD, PhD, Principal Investigator — Johns Hopkins University
Locations (1):
- Johns Hopkins Hospital, Baltimore, Maryland, United States

REFERENCES:
- [Derived] Kho ME, Truong AD, Zanni JM, Ciesla ND, Brower RG, Palmer JB, Needham DM. Neuromuscular electrical stimulation in mechanically ventilated patients: a randomized, sham-controlled pilot trial with blinded outcome assessment. J Crit Care. 2015 Feb;30(1):32-9. doi: 10.1016/j.jcrc.2014.09.014. Epub 2014 Sep 22. PMID 25307979
- [Derived] Kho ME, Truong AD, Brower RG, Palmer JB, Fan E, Zanni JM, Ciesla ND, Feldman DR, Korupolu R, Needham DM. Neuromuscular electrical stimulation for intensive care unit-acquired weakness: protocol and methodological implications for a randomized, sham-controlled, phase II trial. Phys Ther. 2012 Dec;92(12):1564-79. doi: 10.2522/ptj.20110437. Epub 2012 Mar 15. PMID 22421734
- [Derived] Needham DM, Truong AD, Fan E. Technology to enhance physical rehabilitation of critically ill patients. Crit Care Med. 2009 Oct;37(10 Suppl):S436-41. doi: 10.1097/CCM.0b013e3181b6fa29. PMID 20046132

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 3 medical and surgical ICUs at Johns Hopkins Hospitals screened for recruitment from 2008-2009 and 2010-2013 (39 months in total). Recruitment suspended for 17 consecutive months between 2009-2010 due to lack of staffing
Pre-assignment Details: 2 patients (both randomized to the intervention group) were withdrawn PRIOR to any initiation of intervention due to new data arising after randomization (and before intervention initiation) that indicated the subject met the pre-existing exclusion criteria.
Period: Overall Study
Arm/Group | NMES | Sham
Started | 16 | 18
Completed | 12 | 17
Not Completed | 4 | 1
Not completed — Death | 3 | 1
Not completed — encephalopathy; can't do assessment | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | NMES | Sham | Total
Number analyzed (Participants) | 16 | 18 | 34
Age, Continuous [Mean (Standard Deviation); unit: years] | 54 (16) | 56 (18) | 55 (16)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 8 | 17
  Male | 7 | 10 | 17
Region of Enrollment [Number; unit: participants]
  United States | 16 | 18 | 34

OUTCOME MEASURES:

1. Primary Outcome: Lower Extremity Strength, at Hospital Discharge, of 3 Bilateral Muscle Groups (Pretibial, Triceps Surae, and Quadriceps) Measured Via MMT Using a Composite Medical Research Council (MRC) Score
Description: Range 0 to 30 with higher score better. The composite score is a simple sum of the individual scores from the 3 bilateral muscle groups
Time Frame: At hospital discharge
Measure: Mean (Standard Deviation); unit: units (range 0-30; higher is better)
Arm/Group | NMES | Sham
Number analyzed (Participants) | 12 | 17
units (range 0-30; higher is better) | 28 (2) | 27 (3)

2. Secondary Outcome: Individual Muscle Strength Using Handheld Dynamometry: Tibialis Anterior, Gastrocnemius, and Quadriceps Muscle Strength
Description: Strength (in pounds) - measured via handheld dynamometry of tibialis anterior, gastrocnemius, and quadriceps
Time Frame: ICU and hospital discharge
Population: Assessments can only be done on patients who were alive and were able to do participate in the assessment
Measure: Mean (Standard Deviation); unit: pounds
Groups:
- Sham: 60 minute sham sessions every day for the duration of subject's ICU stay. No voltage will be applied to those receiving sham sessions.
  Sham: 60 minute NMES sessions will be applied to three muscle groups of the lower extremities (quadriceps, pretibial, and triceps surae). Sessions start at study entry, and will occur every day for the duration of subject's ICU stay. Sham groups will NOT have voltage applied.
- NMES: 60 minute daily NMES sessions every day for the duration of subject's ICU stay. Neuromuscular Electrostimulation (NMES) CareStim Muscle Stimulation Device (Care Rehab; McLean, VA): 60 minute NMES sessions will be applied to three muscle groups of the lower extremities (quadriceps, pretibial, and triceps surae). Sessions start at study entry, and will occur every day for the duration of subject's ICU stay.
Arm/Group | Sham | NMES
Number analyzed (Participants) | 17 | 12
pounds
  ICU Discharge-tibialis anterior: number analyzed (Participants) | 12 | 8
  ICU Discharge-tibialis anterior | 19 (9) | 21 (10)
  Hospital Discharge-tibialis anterior: number analyzed (Participants) | 12 | 9
  Hospital Discharge-tibialis anterior | 19 (16) | 20 (8)
  ICU Discharge-gastrocnemius: number analyzed (Participants) | 11 | 8
  ICU Discharge-gastrocnemius | 39 (10) | 31 (17)
  Hospital Discharge - gastrocnemius: number analyzed (Participants) | 12 | 9
  Hospital Discharge - gastrocnemius | 31 (14) | 36 (17)
  ICU Discharge - quadriceps: number analyzed (Participants) | 13 | 11
  ICU Discharge - quadriceps | 33 (14) | 28 (14)
  Hospital discharge - quadriceps: number analyzed (Participants) | 15 | 11
  Hospital discharge - quadriceps | 30 (16) | 33 (14)

3. Secondary Outcome: Overall Body Strength
Description: Measuring strength of 6 muscle groups in arms and legs using Medical Research Council composite score (each muscle group scored from scale of 0 [no visible or noticeable contraction] to 5 [maximum strength] and the sum of the scores for the 6 muscle groups equate to a composite score ranging from 0 to 60, higher score is better).
Time Frame: ICU and hospital discharge
Population: Assessments can only be done on patients who were alive and were able to do participate in the assessment
Measure: Mean (Standard Deviation); unit: MRC Composite Score
Arm/Group | NMES | Sham
Number analyzed (Participants) | 12 | 17
MRC Composite Score
  ICU Discharge: number analyzed (Participants) | 12 | 16
  ICU Discharge | 49 (6) | 48 (8)
  Hospital Discharge | 53 (4) | 50 (7)

4. Secondary Outcome: Hand Grip Strength
Description: Hand grip strength measured using a dynamometer (measured in kilograms, then compared to age- and sex-matched population norms to yield % predicted)
Time Frame: ICU and hospital discharge
Population: Assessments can only be done on patients who were alive and were able to do participate in the assessment
Measure: Mean (Standard Deviation); unit: % predicted
Arm/Group | NMES | Sham
Number analyzed (Participants) | 12 | 17
% predicted
  ICU Discharge: number analyzed (Participants) | 12 | 15
  ICU Discharge | 34 (26) | 41 (42)
  Hospital Discharge: number analyzed (Participants) | 12 | 16
  Hospital Discharge | 46 (25) | 40 (28)

5. Secondary Outcome: Respiratory Muscle Strength
Description: Measured using maximal inspiratory pressure (MIP) measurements that is then compared to predicted values for each participant (i.e., % predicted)
Time Frame: ICU and hospital discharge
Population: Assessments can only be done on patients who were alive and were able to do participate in the assessment
Measure: Mean (Standard Deviation); unit: % predicted
Arm/Group | NMES | Sham
Number analyzed (Participants) | 12 | 17
% predicted
  ICU Discharge: number analyzed (Participants) | 3 | 3
  ICU Discharge | 61 (16) | 51 (37)
  Hospital Discharge: number analyzed (Participants) | 3 | 4
  Hospital Discharge | 61 (16) | 51 (37)

6. Secondary Outcome: Functional Status Measured Using Functional Status Score for the Intensive Care Unit
Description: Evaluates a patient's physical function in the ICU setting. Each task is scored, ranging from 0 (unable to perform) to 7 (complete independence).The total score ranges from 0-35, with higher scores indicating better physical functioning.
Time Frame: ICU and hospital discharge
Population: Assessments can only be done on patients who were alive and were able to do participate in the assessment
Measure: Mean (Standard Deviation); unit: FSS-ICU Score
Arm/Group | NMES | Sham
Number analyzed (Participants) | 12 | 17
FSS-ICU Score
  ICU Discharge: number analyzed (Participants) | 12 | 15
  ICU Discharge | 20 (10) | 19 (6)
  Hospital Discharge: number analyzed (Participants) | 12 | 16
  Hospital Discharge | 30 (7) | 26 (8)

7. Secondary Outcome: Duration of Mechanical Ventilation
Description: The number of days the patient was on mechanical ventilation.
Time Frame: Until hospital discharge
Measure: Mean (Standard Deviation); unit: days
Arm/Group | NMES | Sham
Number analyzed (Participants) | 16 | 18
days | 20 (18) | 16 (15)

8. Secondary Outcome: ICU and Hospital Length of Stay
Description: The number of days that the patient was in the ICU and hospital, respectively.
Time Frame: ICU and Hospital discharge
Measure: Mean (Standard Deviation); unit: days
Arm/Group | NMES | Sham
Number analyzed (Participants) | 16 | 18
days
  ICU Length of Stay | 22 (17) | 20 (17)
  Hospital Length of Stay | 36 (22) | 35 (20)

9. Secondary Outcome: ICU and In-hospital Mortality
Description: The number of patients who died in the ICU and those who died by hospital discharge.
Time Frame: ICU discharge and Hospital discharge
Measure: Count of Participants; unit: Participants
Arm/Group | NMES | Sham
Number analyzed (Participants) | 16 | 18
Participants
  ICU Mortality | 3 | 1
  Hospital Mortality | 3 | 3

10. Secondary Outcome: Total Hospital Charges
Description: The total dollar amount of charges from hospital stay
Time Frame: Hospital discharge
Measure: Mean (Standard Deviation); unit: US dollars
Arm/Group | NMES | Sham
Number analyzed (Participants) | 16 | 18
US dollars | 163159 (117730) | 152968 (88683)

11. Secondary Outcome: Hospital Discharge Destination (e.g., Home, Rehab Facility)
Description: Discharge location after hospital stay.
Time Frame: Hospital discharge
Population: Assessments can only be done on patients who were alive and were able to do participate in the assessment
Measure: Count of Participants; unit: Participants
Arm/Group | NMES | Sham
Number analyzed (Participants) | 13 | 15
Participants
  Home | 5 | 8
  Acute rehabilitation | 4 | 6
  Other | 4 | 1

12. Secondary Outcome: Lower Extremity Strength, at Hospital Discharge, of 3 Bilateral Muscle Groups (Pretibial, Triceps Surae, and Quadriceps)
Description: Measured via manual muscle strength test using a composite Medical Research Council (MRC) score with each muscle group rated with score ranging from 0 (no visible or noticeable contraction of the muscle) to 5 (maximum strength). The sum of the scores for the lower limb muscle groups can range from 0 to 30 (higher score is better)
Time Frame: At hospital discharge
Population: Assessments can only be done on patients who were alive and were able to do participate in the assessment
Measure: Mean (Standard Deviation); unit: MRC Score
Arm/Group | NMES | Sham
Number analyzed (Participants) | 12 | 16
MRC Score | 27 (23) | 25 (4)

13. Secondary Outcome: Mean Change in Subject's Lower Extremity Muscle Strength Composite Score From Baseline
Description: The mean change of the sum of the lower limb strength scores between awakening and ICU discharge and between ICU discharge and hospital discharge.
  Three lower limb muscle groups are assessed bilaterally (each muscle group scored from scale of 0 [no visible or noticeable contraction] to 5 [maximum strength]). The scores are then summed for each patient at each time point (range 0 -30, higher score is better).
Time Frame: At ICU and Hospital discharge
Population: Assessments can only be done on patients who were alive and were able to do participate in the assessment
Measure: Mean (Standard Deviation); unit: MRC Score
Arm/Group | NMES | Sham
Number analyzed (Participants) | 16 | 18
MRC Score
  Awakening to ICU Discharge: number analyzed (Participants) | 10 | 11
  Awakening to ICU Discharge | 5.3 (5.9) | 0.8 (3.8)
  ICU Discharge to Hospital Discharge: number analyzed (Participants) | 12 | 15
  ICU Discharge to Hospital Discharge | 5.7 (5.1) | 1.8 (2.7)

14. Secondary Outcome: ICU Delirium
Description: Proportion of ICU days the patient had delirium
Time Frame: During ICU stay - on days with study (NMES/Sham) session
Measure: Mean (Standard Deviation); unit: Mean % delirious days
Units Other Than Participants: Days of session
Arm/Group | NMES | Sham
Number analyzed (Participants) | 16 | 18
Number analyzed (Days of session) | 106 | 172
Mean % delirious days | 67 (34) | 66 (32)

15. Secondary Outcome: Subgroup Analysis
Description: For patients with >= 7 days of mechanical ventilation, we will compare the 2 groups for the following outcomes: Lower extremity muscle strength, mean change in whole body muscle strength score from baseline to ICU discharge, mean change in whole body muscle strength score from baseline to hospital discharge, and whole body muscle strength score at ICU discharge and at hospital discharge.
  Each muscle group is assessed bilaterally (scale of 0 [no visible or noticeable contraction] to 5 [maximum strength]). There are three muscle groups assessed bilaterally for lower extremity (hip flexion, knee extension, and ankle dorsiflexion) (score range 0-30, higher score is better i.e. stronger); while for whole body strength assessment (score range 0-360, higher score is better), the following additional muscles are assessed: shoulder abduction, elbow flexion and wrist extension.
  The scores are then summed for each patient at each time point.
Time Frame: ICU and hospital discharge and change over time
Population: This was an a priori subgroup analyses of patients who had mechanical ventilation duration >=7 days. Not all participants could be evaluated at each time point (e.g. cognitive status) and this explains the different sample sizes for each outcome.
Measure: Mean (Standard Deviation); unit: muscle strength score (higher is better)
Arm/Group | NMES | Sham
Number analyzed (Participants) | 11 | 14
muscle strength score (higher is better)
  Lower extremity muscle strength at ICU discharge: number analyzed (Participants) | 11 | 13
  Lower extremity muscle strength at ICU discharge | 27 (2) | 25 (4)
  Lower extremity muscle strength at hospital discha | 28 (2) | 27 (3)
  Whole body muscle strength score at ICU discharge: number analyzed (Participants) | 11 | 13
  Whole body muscle strength score at ICU discharge | 48 (6) | 48 (8)
  Whole body muscle strength score at hospital disch | 53 (4) | 50 (7)
  Mean change in whole body strength (bsln to ICU): number analyzed (Participants) | 9 | 8
  Mean change in whole body strength (bsln to ICU) | 7.9 (8.8) | 3.4 (5.7)
  Mean change-whole body strength (bsln to hosp. dc): number analyzed (Participants) | 11 | 12
  Mean change-whole body strength (bsln to hosp. dc) | 11.6 (8.9) | 5.8 (5.4)

ADVERSE EVENTS:
Arm/Group | NMES | Sham
Serious Adverse Events (participants affected / at risk) | 0/16 | 0/18
Other Adverse Events (participants affected / at risk) | 0/16 | 0/18

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No